CLINICAL TRIAL: NCT00985283
Title: Feasibility and Effects of Preventive Home Visits for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21-AG29502-2; R21-AG29502-2; R21AG029502 (NIH)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Frailty
Keywords: prevention; older adults; function; participation; life satisfaction; self-rated health
MeSH Terms: conditions — Frailty; Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preventive home visit (Experimental): receives preventive home visit intervention 4 times over 1 year
  Interventions: Behavioral: Preventive home visit
- comparison group (Active Comparator): receives information packets on local services for older adults and health promotion material twice during 1 year
  Interventions: Behavioral: minimal intervention

INTERVENTIONS:
Behavioral: Preventive home visit — in-home visit by a trained occupational therapist to assess older adult's living context and occupational performance and to provide recommendations for changes or continuation of behavior or context
  Arms: Preventive home visit
Behavioral: minimal intervention — provision of information related to services and health promotion for older adults as a low-cost minimal alternative to the intervention
  Arms: comparison group

SUMMARY:
The goals of this project are to implement an innovative intervention for older adults and assess both its feasibility and effects on health and well-being. The investigators hypothesize that the intervention group will show a significantly better slope for a range of outcomes during and after the intervention.

DETAILED DESCRIPTION:
Aging in place is now recognized as a goal of most older adults. While medically driven interventions such as home health care assist older adults to age in place, these occur not as true preventive measures but as reactions to losses in function or health. The search for preventive methods to mitigate decline and unwanted moves from home and community is important. One such method, Preventive Home Visits (PHVs), has been utilized in parts of Europe for approximately two decades. The PHV model is based on infrequent but regular visits to an older adult's home by a trained practitioner (typically an occupational therapist or nurse). The visit is designed to assess the older person's situation and provide information and advice to optimize function and well-being. Evidence about PHV efficacy is mixed but generally supportive, and there is a distinct need to create and examine a preventive non-medical intervention model in the USA. A successfully developed and implemented approach could enhance lives and save costs. We plan to implement an intervention informed by a framework based on a synthesis of the World Health Organization function and disability model and the Occupational Therapy Practice Framework. We aim to implement and evaluate this PHV intervention in Orange County, North Carolina to assess the feasibility and effects of preventive home visits with older adults. We will use an experimental, repeated measures design in which approximately 120 older (75+ years) community-dwelling adults who are at-risk for functional decline are randomly assigned to experimental and comparison groups. The experimental group will receive the PHV intervention four times across a 12 month period. The comparison group will receive a minimal intervention of two informational phone calls and printed materials about local services during the same period. An occupational therapist with the requisite training and experience in home-based evaluation and intervention will conduct the experimental intervention. We will independently administer a set of standardized scales to both groups immediately pre-intervention, and again at regular intervals after each intervention. These outcome measures will cover the primary dimensions on which we hypothesize PHVs will have a positive influence: functional ability, participation, self-efficacy, life satisfaction, and self-reported health. Secondary outcomes include hospitalization and institutionalization. Analyses will compare the differences in outcomes for the two groups as well as assess several dimensions of intervention feasibility. These data will be the basis for a subsequent, enhanced intervention and study.

ELIGIBILITY:
Inclusion Criteria:

* 75 years or older
* lives in community (not in nursing home or assisted living)
* not currently receiving home health services
* vulnerable elders survey score of 3 or higher

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
functional ability | 5 times across approx. 15 months

SECONDARY OUTCOMES:
life satisfaction | 5 times across approx. 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm P. Cutchin, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Cutchin MP, Coppola S, Talley V, Svihula J, Catellier D, Shank KH. Feasibility and effects of preventive home visits for at-risk older people: design of a randomized controlled trial. BMC Geriatr. 2009 Dec 3;9:54. doi: 10.1186/1471-2318-9-54. PMID 19958547